CLINICAL TRIAL: NCT03596541
Title: Clinical Validation of Tele-stethoscope System Digital Bluetooth Ehas-fundatel
Brief Title: Clinical Validation of Tele-stethoscope System Digital
Acronym: TeleCáceres
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Jaime Corral Penafiel, medical doctor, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: T-stethoscopy
Record Dates: First submitted 2014-06-16; First posted 2018-07-24 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Disorder; Heart Disorder
Keywords: Telemedicina; Respiratory sounds; Tele-stethoscopy; Wireless; Real-time; e-health; Heart sounds
MeSH Terms: conditions — Respiration Disorders; Heart Diseases; Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- An open real-time tele-stethoscopy system (Experimental): EHAS-Fundatel digital stethoscope is an open real-time tele-stethoscopy system. The interventions in this arm will be to make a respiratory and heart auscultation with this tele-stethoscope. After that, we will do the comparison or agreetment between the auscultation of two protocols: tele-stethoscopy system and conventional stethoscope.
  Interventions: Device: Heart and Respiratory Auscultation of an open real-time tele-stethoscopy system (EHAS-Fundatel digital stethoscope)
- Conventional stethoscope (Active Comparator): Conventional stethoscope used is the 3M Littmann Classic II S.E. stethoscope. The interventions in this arm will be to make a respiratory and heart auscultation with this conventional stethoscope. After that we will do the comparison or agreetment between the ascultation of two protocols: conventional stethoscope and tele-stethoscopy system.
  Interventions: Device: Heart and Respiratory Auscultation of an open real-time tele-stethoscopy system (EHAS-Fundatel digital stethoscope)

INTERVENTIONS:
Device: Heart and Respiratory Auscultation of an open real-time tele-stethoscopy system (EHAS-Fundatel digital stethoscope) — We compare the respiratory and heart auscultation of clinicians using the EHAS-Fundatel digital stethoscope and a conventional stethoscope and we will observe; inter-observer and intra-observer differences by two auscultation methods.

SUMMARY:
Acute respiratory infections and other respiratory and cardiology diseases like COPD or heart failure are important causes of morbidity and mortality around the world. Telemedicine is defined as the delivery of health care and the sharing of medical knoledge over distances using telecommunication systems. Inexpensive techologies offer the possibility of a direct, real-time connection between the patient or the other end. These technologies help to the physicians to manage different symptoms and cardio-respiratory diseases. A real-time wireless tele-stethoscopy system was designed to allow a physician to receive real-time cardio-respiratory sounds from a remote auscultation, as well as video images showing where the technician is placing the stethoscope on the patient´s body. Actually, the lack of physicians in rural areas of developing countries makes difficult their correct diagnosis and treatment. Furthermore, in the majority of health systems, the patients are shared between primary care and medical specialty in hospitals. The tele-stethoscopy system through telemedicine could help to the physicians or health-care technicians in the majority of health systems and especially in rural areas of developing countries without physicians to manage the patients. For this reason, the goal of this project is the clinical validation of an open real-time tele-stethoscope systme (EHAS-Fundatel digital stethoscope) previously designed, with different specialist (pneumologists, cardiologists and internists.)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent sign.
* Pacient admitted to hospital with any disease but no inestable disease.

Exclusion Criteria:

* The lack of informed consent.
* Inestable disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2018-11-27 (Actual); Study Completion 2018-12-27 (Actual)

PRIMARY OUTCOMES:
Intra-observer agreement for heart murmurs auscultation using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will randomize the first auscultation (baseline auscultation) into tele-stethoscope system or conventional stethoscope. After 1 hour, we will use the other auscultation method.
  The investigators will measure if there is a heart murmur or not and the intra-observer agreement by the kappa index in the heart murmurs auscultation.
Intra-observer agreement for heart rhythm auscultation using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will measure if there is a heart rhythm auscultation or not rhythm and the intra-observer agreement by the kappa index in the heart rhythm auscultation.
Intra-observer agreement for vesicular murmur auscultation using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will measure if there is a normal vesicular murmur or not and the intra-observer agreement by the kappa index in the vesicular murmur auscultation.
Intra-observer agreement for lung rales sounds using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will measure if there is a lung rale sound or not and the intra-observer agreement by the kappa index in the lung rale sound.

SECONDARY OUTCOMES:
Inter-observer agreement for for heart murmurs auscultation using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will randomize the first auscultation (baseline auscultation) into tele-stethoscope system or conventional stethoscope. After 1 hour, we will use the other auscultation method.
  The investigators will measure if there is a heart murmur or not and the inter-observer agreement by the kappa index in the heart murmurs auscultation.
Inter-observer agreement for heart rhythm auscultation using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will measure if there is a heart rhythm auscultation or not rhythm and the inter-observer agreement by the kappa index in the heart rhythm auscultation.
Inter-observer agreement for vesicular murmur auscultation using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will measure if there is a normal vesicular murmur or not and the inter-observer agreement by the kappa index in the vesicular murmur auscultation.
Inter-observer agreement for lung rales sounds using the two methods (tele-stethoscope and conventional stethoscope) | change from baseline auscultation to final auscultation (after 1 hour)
  The investigators will measure if there is a lung rale sound or not and the inter-observer agreement by the kappa index in the lung rale sound.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Corral, MD, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- San Pedro de Alcántara Hospital, Cáceres, Spain